CLINICAL TRIAL: NCT02717377
Title: Effect of Frequent Interruptions of Prolonged Sitting on Self-perceived Levels of Energy, Mood, Food Cravings and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13-2777
Record Dates: First submitted 2016-02-22; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Mood; Energy; Food Cravings; Cognitive Function
Keywords: Micro bouts; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Uninterrupted sitting (No Intervention): Subjects remained seated all day except to rise from the chair to void.
- Sitting + one bout of activity (Active Comparator): Subjects remained seated all day, except to rise from the chair to void, and to perform one bout of 30-minutes moderate-intensity walking. Physical activity was performed at 0800, after measures of vitals and basal questionnaire assessments, but before breakfast.
  Interventions: Behavioral: physical activity
- Sitting + microbursts of activity (Experimental): Subjects rose from the seated position every hour for 6-hours from 0910 to 1430 to complete 5-minute bouts of moderate-intensity walking, yielding a total activity time of 30-minutes.
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity
  Arms: Sitting + microbursts of activity; Sitting + one bout of activity

SUMMARY:
This study is designed to test the effects of six 5 minute microbursts of physical activity spread across the day as compared to either a sedentary control condition or a single 30 minute bout of moderate intensity physical activity on cognitive function, self-reported energy levels, aspects of eating behavior and measures of metabolic health. The primary hypotheses are:

1. Hourly 5 minute bouts of moderate intensity exercise during the day will increase afternoon cognitive function as compared to a no exercise condition.
2. Hourly 5 minute bouts of moderate intensity exercise during the day will increase afternoon cognitive function more than a single 30 minute AM bout.

Secondary exploratory hypotheses include

1. Hourly 5 minute bouts of moderate intensity exercise during the day will increase self-reported energy levels, reduce orexigenic appetitive measures and improve measures of metabolic health as compared to a no exercise condition.
2. Hourly 5 minute bouts of moderate intensity exercise during the day will increase self-reported energy levels, reduce orexigenic appetitive measures and improve measures of metabolic health more than a single 30 minute AM bout.

ELIGIBILITY:
Inclusion Criteria:

1. All ethnic groups and both genders
2. Age: Lower age limit: 19 years; Upper age limit: 45 years
3. Body-mass Index: Lower BMI limit: 18.5 kg/m2; Upper BMI limit: 29.9 kg/m2
4. Willing to adhere to caffeine restrictions of no more than two 16 ounce beverages in the morning of each study day with no caffeine intake after 12:00pm on any of the three study days

Exclusion Criteria:

1. History of cardiovascular disease, including coronary artery disease, congestive heart failure, & unstable angina, or uncontrolled hypertension (>140/90 mm Hg)
2. Currently smoking or stopped smoking in the last 6 months
3. Medications affecting weight, energy intake, or energy expenditure in the last 6 months
4. Use of oral steroids
5. History of stroke or seizures, thyroid disease, type 1 or 2 diabetes, Cushing's syndrome, cerebrovascular, renal disease, hepatic disease, arrhythmias
6. Cancer requiring treatment in the past 5 years, with the exception of skin cancers other than melanoma
7. Infectious diseases: Self-reported HIV positivity or active tuberculosis
8. Inability to exercise for more than 30 minutes on a treadmill at moderate intensity
9. Currently pregnant, lactating or less than 6 months post-partum
10. History of a major psychiatric disorder including schizophrenia, bipolar illness or psychotic depression
11. Score of >25 on Beck Depression Inventory
12. No recreational drug use including marijuana in the past 1 year

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Energy and Mood level | During each of the three separate study days energy and mood levels are assessed at (in minutes): T0, T40, T70, T80, T90, T120, T140, T230, T350, T390, T400, T405, T410, and T435
  Self-perceived energy and mood were measured by using visual analogue scales (VAS) as described below at baseline.
Change in Cognitive function | During each of the three separate study days cognitive function is measured at (in minutes): T410
  The flanker task is used to measure cognitive function
Change in Cognitive Function | During each of the three separate study days cognitive function is measured at (in minutes): T425
  After the Flanker task, the Comprehensive Trail Making Test is used to measure cognitive function during each study day.

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
This clinical trial is a small study (n=30) that received limited funding from Johnson and Johnson Company, a non-public funding company. Our data sharing plan will follow the NIH guidelines for data sharing plans of small clinical trials and not unique set of data that could benefit the community (http://grants.nih.gov/grants/policy/data_sharing/data_sharing_faqs.htm#901). Following the NIH definition of "the timely release and sharing" to be no later than the acceptance for publication of the main findings from the final data set, final research data will be shared through scientific publications after peer-review.

REFERENCES:
- [Derived] Bergouignan A, Legget KT, De Jong N, Kealey E, Nikolovski J, Groppel JL, Jordan C, O'Day R, Hill JO, Bessesen DH. Effect of frequent interruptions of prolonged sitting on self-perceived levels of energy, mood, food cravings and cognitive function. Int J Behav Nutr Phys Act. 2016 Nov 3;13(1):113. doi: 10.1186/s12966-016-0437-z. PMID 27809874